CLINICAL TRIAL: NCT02956616
Title: Enhanced Recovery at Cesarean Birth to Improve Postoperative Outcomes and Reduce Postoperative Length of Stay
Acronym: ERAC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Peter S. Bernstein, Principal Investigator, Montefiore Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2016-6966
Record Dates: First submitted 2016-11-02; First posted 2016-11-07 (Estimated); Results first posted 2019-04-25 (Actual); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Cesarean Section
Keywords: Enhanced Recovery
MeSH Terms: interventions — Ketorolac; Ketorolac Tromethamine; Chewing Gum; Xylitol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Enhanced Recovery (Experimental): Postoperative recovery will follow the usual service protocols as if the patient were not in the study with the exception of components of the enhanced recovery protocol (detailed previously), which will include several evidence-based recommendations including early ambulation, early diet initiation, early removal of urinary catheter, early removal of postoperative dressing. Additionally, participants in this group will receive intravenous ketorolac for pain control and Xylitol chewing gum for improvement of postoperative gastrointestinal function.
  Interventions: Drug: ketorolac; Other: Chewing Gum; Procedure: Enhanced Recovery Protocol
- Routine Perioperative Care (Active Comparator): Postoperative recovery will follow the usual service protocols at our institution. Participants in this group may receive intravenous ketorolac (toradol) for pain control
  Interventions: Drug: ketorolac

INTERVENTIONS:
Drug: ketorolac — Ketorolac, sold under the brand name Toradol among others, is a nonsteroidal anti-inflammatory drug in the family of heterocyclic acetic acid derivatives, used as an analgesic. It is considered a first-generation NSAID. Ketorolac acts by inhibiting the bodily synthesis of prostaglandins.
  Other Names: Toradol
Other: Chewing Gum — Xylitol chewing gum will be provided to patients immediately after the procedure and will be provided 3 times per day for a duration of 30 minutes at each time, based on a metanalysis and systematic review. Patient's will be encouraged on its use for return of bowel function.
  Other Names: Xylitol
  Arms: Enhanced Recovery
Procedure: Enhanced Recovery Protocol — enhanced recovery protocol (detailed previously) will include several evidence-based recommendations including early ambulation, early diet initiation, early removal of urinary catheter, early removal of postoperative dressing and standing ketorolac for 24 hours postoperatively.
  Arms: Enhanced Recovery

SUMMARY:
To determine whether women randomized to an enhanced recovery program will have improved postoperative outcomes including improved breastfeeding initiation and continuation, reduction in hospital length of stay without compromising patient satisfaction in comparison to standard postoperative recovery interventions.

DETAILED DESCRIPTION:
The investigators hypothesize that an enhanced recovery program which includes several evidence based interventions at the time of cesarean birth in obstetrics will promote early ambulation, resumption of diet and initiation of breastfeeding, and reduce postoperative hospital length of stay.

Enhanced Recovery Protocol Components:

1. Provide preoperative education about the perioperative recovery experience including postoperative analgesia, thromboprophylaxis and breastfeeding education
2. Minimize preoperative starvation times

   1. Moderate amount of clears up to 2 hours prior to anesthesia
   2. Solid foods up to 6-8 hours prior to anesthesia
3. Prophylactic antibiotics
4. Venous thromboembolism prophylaxis (mechanical) initiated at the time of cesarean birth and continued postoperatively
5. Chewing gum (Xylitol) to reduce postoperative ileus
6. Routine administration of Non-steroidal anti-inflammatory drug, Ketorolac, 15mg every hour for 24 hours postoperatively to minimize postoperative narcotic use
7. Early initiation of feeding after cesarean, immediately for clears, 30 minutes for regular diet as tolerated
8. Early removal of urinary catheter (12 hours postoperatively)
9. Early removal of dressing (6 hours postoperatively)
10. Early mobilization at 12 hours after delivery
11. Early skin-to- skin/breastfeeding initiation
12. Early incentive spirometry

Currently, patients are encouraged to ambulate on the first post-operative day, but it is largely left up to the patient when to actually begin to ambulate. They are similarly offered a diet on the first postoperative day but are not encouraged to eat. Breastfeeding is more systematically encouraged early as part of Montefiore's effort to get baby friendly designation. And finally, patients are typically discharged on postoperative day number three unless complications arise in the newborn or the mother. As part of this study, patients in both the enhanced recovery and usual care group will be offered the opportunity to be discharged from the hospital on postoperative day number 2 if their recovery is progressing well and if they choose not to leave then they will be encouraged to return home on postoperative day number 3 according to the current standard of care.

ELIGIBILITY:
Inclusion Criteria:

1. Women undergoing a non-urgent or elective cesarean delivery >37 weeks gestation

Exclusion Criteria:

1. Women undergoing an urgent or emergent cesarean birth
2. Women less than 18 years old
3. Patients receiving general anesthesia
4. Abnormally adherent placenta (Placenta Accreta) or expected excessive blood loss (Placenta accreta)
5. Pre-existing essential hypertension or hypertensive disorders of pregnancy (preeclampsia, eclampsia, HELLP)
6. Chronic or acute renal impairment
7. Bleeding disorders or platelet dysfunction
8. Peptic ulcer disease or gastrointestinal bleeding
9. Known hypersensitivity to ketorolac (toradol)
10. Active infection at the time of cesarean
11. Cesarean birth prior to 37 weeks
12. Women in significant pain in labor

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-06-15 (Actual); Study Completion 2018-06-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wrench IJ, Allison A, Galimberti A, Radley S, Wilson MJ. Introduction of enhanced recovery for elective caesarean section enabling next day discharge: a tertiary centre experience. Int J Obstet Anesth. 2015 May;24(2):124-30. doi: 10.1016/j.ijoa.2015.01.003. Epub 2015 Jan 14. PMID 25794417
- [Background] Brooten D, Roncoli M, Finkler S, Arnold L, Cohen A, Mennuti M. A randomized trial of early hospital discharge and home follow-up of women having cesarean birth. Obstet Gynecol. 1994 Nov;84(5):832-8. PMID 7936522
- [Background] Practice Guidelines for Obstetric Anesthesia: An Updated Report by the American Society of Anesthesiologists Task Force on Obstetric Anesthesia and the Society for Obstetric Anesthesia and Perinatology. Anesthesiology. 2016 Feb;124(2):270-300. doi: 10.1097/ALN.0000000000000935. No abstract available. PMID 26580836
- [Background] Habib AS, George RB, McKeen DM, White WD, Ituk US, Megalla SA, Allen TK. Antiemetics added to phenylephrine infusion during cesarean delivery: a randomized controlled trial. Obstet Gynecol. 2013 Mar;121(3):615-623. doi: 10.1097/AOG.0b013e3182839fee. PMID 23635626
- [Background] Masood SN, Masood Y, Naim U, Masood MF. A randomized comparative trial of early initiation of oral maternal feeding versus conventional oral feeding after cesarean delivery. Int J Gynaecol Obstet. 2014 Aug;126(2):115-9. doi: 10.1016/j.ijgo.2014.02.023. Epub 2014 Apr 29. PMID 24856433
- [Background] Huang H, Wang H, He M. Early oral feeding compared with delayed oral feeding after cesarean section: a meta-analysis. J Matern Fetal Neonatal Med. 2016;29(3):423-9. doi: 10.3109/14767058.2014.1002765. Epub 2015 Mar 10. PMID 25754213
- [Background] Guo J, Long S, Li H, Luo J, Han D, He T. Early versus delayed oral feeding for patients after cesarean. Int J Gynaecol Obstet. 2015 Feb;128(2):100-5. doi: 10.1016/j.ijgo.2014.07.039. Epub 2014 Oct 22. PMID 25457588
- [Background] Saad AF, Saoud F, Diken ZM, Hegde S, Kuhlmann MJ, Wen TS, Hankins GD, Saade GR, Costantine MM. Early versus Late Feeding after Cesarean Delivery: A Randomized Controlled Trial. Am J Perinatol. 2016 Mar;33(4):415-9. doi: 10.1055/s-0035-1565918. Epub 2015 Oct 19. PMID 26479169
- [Background] Craciunas L, Sajid MS, Ahmed AS. Chewing gum in preventing postoperative ileus in women undergoing caesarean section: a systematic review and meta-analysis of randomised controlled trials. BJOG. 2014 Jun;121(7):793-9; discussion 799. doi: 10.1111/1471-0528.12696. Epub 2014 Mar 14. PMID 24628729
- [Background] Zhu YP, Wang WJ, Zhang SL, Dai B, Ye DW. Effects of gum chewing on postoperative bowel motility after caesarean section: a meta-analysis of randomised controlled trials. BJOG. 2014 Jun;121(7):787-92. doi: 10.1111/1471-0528.12662. Epub 2014 Mar 14. PMID 24629205
- [Background] Shang H, Yang Y, Tong X, Zhang L, Fang A, Hong L. Gum chewing slightly enhances early recovery from postoperative ileus after cesarean section: results of a prospective, randomized, controlled trial. Am J Perinatol. 2010 May;27(5):387-91. doi: 10.1055/s-0029-1243313. Epub 2009 Dec 11. PMID 20013603
- [Background] Peleg D, Eberstark E, Warsof SL, Cohen N, Ben Shachar I. Early wound dressing removal after scheduled cesarean delivery: a randomized controlled trial. Am J Obstet Gynecol. 2016 Sep;215(3):388.e1-5. doi: 10.1016/j.ajog.2016.03.035. Epub 2016 Mar 25. PMID 27018465
- [Background] Lowder JL, Shackelford DP, Holbert D, Beste TM. A randomized, controlled trial to compare ketorolac tromethamine versus placebo after cesarean section to reduce pain and narcotic usage. Am J Obstet Gynecol. 2003 Dec;189(6):1559-62; discussion 1562. doi: 10.1016/j.ajog.2003.08.014. PMID 14710063
- [Background] El-Mazny A, El-Sharkawy M, Hassan A. A prospective randomized clinical trial comparing immediate versus delayed removal of urinary catheter following elective cesarean section. Eur J Obstet Gynecol Reprod Biol. 2014 Oct;181:111-4. doi: 10.1016/j.ejogrb.2014.07.034. Epub 2014 Aug 1. PMID 25145762
- [Result] Adamina M, Kehlet H, Tomlinson GA, Senagore AJ, Delaney CP. Enhanced recovery pathways optimize health outcomes and resource utilization: a meta-analysis of randomized controlled trials in colorectal surgery. Surgery. 2011 Jun;149(6):830-40. doi: 10.1016/j.surg.2010.11.003. Epub 2011 Jan 14. PMID 21236454
- [Derived] Teigen NC, Sahasrabudhe N, Doulaveris G, Xie X, Negassa A, Bernstein J, Bernstein PS. Enhanced recovery after surgery at cesarean delivery to reduce postoperative length of stay: a randomized controlled trial. Am J Obstet Gynecol. 2020 Apr;222(4):372.e1-372.e10. doi: 10.1016/j.ajog.2019.10.009. Epub 2019 Oct 26. PMID 31669738

RESULTS

PARTICIPANT FLOW:
Groups:
- Enhanced Recovery: Postoperative recovery will follow the usual service protocols as if the patient were not in the study with the exception of components of the enhanced recovery protocol (detailed previously), which will include several evidence-based recommendations including early ambulation, early diet initiation, early removal of urinary catheter, early removal of postoperative dressing. Additionally, participants in this group will receive intravenous ketorolac for pain control and Xylitol chewing gum for improvement of postoperative gastrointestinal function.
  ketorolac: Ketorolac, sold under the brand name Toradol among others, is a nonsteroidal anti-inflammatory drug in the family of heterocyclic acetic acid derivatives, used as an analgesic. It is considered a first-generation NSAID. Ketorolac acts by inhibiting the bodily synthesis of prostaglandins.
  Chewing Gum: Xylitol chewing gum will be provided to patients immediately after the procedure and will be provided 3 times per day for
Period: Overall Study
Arm/Group | Enhanced Recovery | Routine Perioperative Care
Started | 58 | 60
Completed | 58 | 60
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Enhanced Recovery | Routine Perioperative Care | Total
Number analyzed (Participants) | 58 | 60 | 118
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 58 | 60 | 118
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.43 (4.92) | 31.93 (5.43) | 31.18 (5.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 60 | 118
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 4 | 4 | 8
  African American | 13 | 16 | 29
  Hispanic | 33 | 29 | 62
  Asian | 3 | 2 | 5
  Other | 5 | 9 | 14

OUTCOME MEASURES:

1. Primary Outcome: Discharge on Postoperative Day #2
Description: Number of patients discharged on postoperative Day #2
Time Frame: Until patient's day of hospital discharge or a maximum of one month from cesarean delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced Recovery | Routine Perioperative Care
Number analyzed (Participants) | 58 | 60
Participants | 5 | 2

2. Secondary Outcome: Postoperative Pain Medication Requirement
Description: The amount of postoperative pain medication required for each patient in Morphine Milligram Equivalents
Time Frame: Until patient's day of hospital discharge or a maximum of one month from cesarean delivery
Measure: Mean (Standard Deviation); unit: Morphine Milligram Equivalents
Arm/Group | Enhanced Recovery | Routine Perioperative Care
Number analyzed (Participants) | 58 | 60
Morphine Milligram Equivalents | 117.16 (54.17) | 119.38 (47.98)

3. Secondary Outcome: Breastfeeding Initiation
Description: All patients will be queried regarding whether breastfeeding was initiated after cesarean birth and how soon after birth
Time Frame: Until patient's day of hospital discharge or a maximum of one month from cesarean delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced Recovery | Routine Perioperative Care
Number analyzed (Participants) | 58 | 60
Participants
  Breastfeeding | 39 | 29
  Bottlefeeding | 4 | 2
  Both Breastfeeding and Bottlefeeding | 15 | 29

4. Secondary Outcome: Postoperative Length of Hospital Stay
Description: Postoperative Length of Hospital Stay in Hours from time of surgery
Time Frame: Until patient's day of hospital discharge or a maximum of one month from cesarean delivery
Measure: Median (Inter-Quartile Range); unit: Hours
Arm/Group | Enhanced Recovery | Routine Perioperative Care
Number analyzed (Participants) | 58 | 60
Hours | 73.58 [71.08 to 76.62] | 75.50 [72.86 to 76.84]

ADVERSE EVENTS:
Time Frame: Throughout the duration of study from enrollment until 6 weeks after surgery
Arm/Group | Enhanced Recovery | Routine Perioperative Care
All-Cause Mortality (participants affected / at risk) | 0/58 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/58 | 0/60
Other Adverse Events (participants affected / at risk) | 0/58 | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-05): https://cdn.clinicaltrials.gov/large-docs/16/NCT02956616/Prot_SAP_000.pdf